CLINICAL TRIAL: NCT05385679
Title: Comparison of Two Flaps in Surgical Removal of Impacted Lower Third Molar;a Randomized Comparative Double Blind Study
Brief Title: Comparison of Two Flaps in Surgical Removal of Impacted Lower Third Molar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ashutosh Kumar Singh (Other)
Responsible Party: Sponsor-Investigator, Ashutosh Kumar Singh, Lecturer of department Oral And Maxillofacial Surgery, College of Medical Sciences Teaching Hospital. Nepal
Organization: College of Medical Sciences Teaching Hospital. Nepal (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOM2
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envelop Flap (Active Comparator): An envelope flap designs involves a sulcular incision from the first to the second molar and a distal relieving incision to the mandibular ramus.
  Interventions: Procedure: Surgical Extraction of lower third molar
- Triangular flap (Active Comparator): Triangular flap involves incision from the mandibular ramus to the distobuccal crown edge of the second molar, followed by a perpendicular incision obliquely into the mandibular vestibulum, with a length of about 10 mm.
  Interventions: Procedure: Surgical Extraction of lower third molar

INTERVENTIONS:
Procedure: Surgical Extraction of lower third molar — The surgical removal of mandibular third molar is one of the most common procedures done in oral and maxillofacial surgery. Patients often experience pain, swelling, trismus, dehiscence, alveolar osteitis, infection, nerve injury and periodontal tissue damage after third molar surgery. Flap design is an important step in third molar surgery. Envelope flap and modifications of triangular flap are the two most commonly used flaps in surgical removal of lower third molar.

SUMMARY:
Project summary

The surgical removal of mandibular third molar is one of the most common procedures done in oral and maxillofacial surgery. Patients often experience pain, swelling, trismus, dehiscence, alveolar osteitis, infection, nerve injury and periodontal tissue damage after third molar surgery. Flap design is an important step in third molar surgery.The aim of this study is to compare the triangular and envelope flap designs in lower third molar surgery in terms of postoperative sequelae including pain ,trismus,swelling,incidence of dry socket and also operative time taken.The study also aims to find out does the level of impacted mandibular third molar and number of roots has effect on postoperative outcomes in surgical removal of mandibular third molar.The study design used will be a double-blind randomized clinical study. Patients who fit the inclusion criteria will be included as research subjects.Sample will be divided into two groups randomly. In one group the envelope flap will be raised during surgical removal of the lower third molar while in the other triangular flap will be used.

Investigators will also divide the third molars into level 1,level 2,level 3 based on the relationship between the tip of mesial cusp of impacted third molar and the distal surface of crown of adjacent second molar based on orthopantomograph findings.Level 1 will be when the tip of mesial cusp of third molar is within the occlusal third of crown of second molar,level 2 will be when the tip of mesial cusp of third molar is within the middle third of crown of second molar, level 3 will be when the tip of mesial cusp of third molar is within and below the cervical third of crown of second molar.

Another subgroup will be based on the number of roots of the impacted third molar where investigators will divide the third molar into single rooted and multirooted based on orthopantomograph findings.

Investigators will also divide the sample based on gender and age group as below 30 years and above 30 years.

The primary outcomes to be measured are pain and operative time while secondary outcomes are swelling ,trismus and incidence of dry socket.Outcome assessment will be done by another clinician than surgeon using scientific tools and techniques as mentioned.

Surgical procedures and outcomes measurement will be done by separate clinicians to ensure masking.

DETAILED DESCRIPTION:
Andreasen et al (1997) defines impaction as a cessation of the eruption of a tooth caused by a clinically or radiographically detectable physical barrier in the eruption path or by an ectopic position of the tooth. The prevalence of third molar impaction ranges from 16.7% to 68.6%. Common pathologies associated with third molars are pericoronitis, caries of impacted teeth or adjacent tooth, second molar tooth resorption, periodontal bone loss of adjacent tooth and odontogenic cysts. The surgical removal of mandibular third molar is one of the most common procedures done in oral and maxillofacial surgery. Flap design is an important step in third molar surgery.Commonly used flap in surgical removal of third molar are envelope flap and triangular flap with modifications.

A number of classifications have been developed for impacted third molars.The most widely used are;

1. Angulation (Winter, 1926) of the impacted tooth ; Vertical, Mesioangular, Horizontal, Distoangular
2. Relationship of the impacted tooth to the anterior border of the ramus (Pell and Gregory, 1942); Class I: Sufficient space available anterior to the anterior border of ramus for the third molar to erupt.

   Class II: Space available is less than the mesio distal width of the crown of the third molar Class III: All or most of the third molar is located within the ramus.
3. Depth of impaction (Pell and Gregory Classification based on relationship to occlusal plane); Position A: The highest portion of the tooth (occlusal plane) is on a level with or above the occlusal line.

Position B: The highest portion of the tooth is below the occlusal line but above the cervical line of the second molar.

Position C: The highest portion of the tooth is below the cervical line of the second molar.

Rationale and justifications of study

The surgical removal of mandibular third molar is one of the most common procedure done in oral and maxillofacial surgery and often associated with pain, swelling, trismus, dehiscence, alveolar osteitis, infection, nerve injury and periodontal tissue damage.Flap design is an important step in this procedure.

The present study is aimed at comparing the envelope and triangular flap in lower third molar surgery based on postoperative outcomes.The study also aims to find does the number of roots and also the relation between level of mesial cusp tip of impacted lower third molar and distal surface of adjacent second molar has any effect on postoperative sequelae.

Although much research was done so far on this topic,further studies were suggested .

Both envelope and triangular flaps are routinely used in lower third molar surgery.So,this study claims no extra medical risks related to the intervention.Patients and investigators bear no extra economic burden in investigations and research.

Objectives

General:

To compare the triangular and envelope flap in surgical removal of vertical and mesioangular impacted lower third molar.

Specific:

To evaluate whether the relation between level of mesial cusp tip of impacted third molar to the distal surface of adjacent second molar has any effect on the post operative outcomes independent of flap designs.

To evaluate the effect of the number of roots of impacted third molar to the postoperative outcomes in third molar surgery independent of flap designs.

Research hypothesis

Null hypothesis: There is no difference between the envelope and triangular flap in terms of post operative outcomes in surgical removal of vertical and mesioangular impacted mandibular third molar.

Alternate hypothesis:There is significant difference between envelope and triangular flap in terms of post operative outcomes in surgical removal of vertical and mesioangular impacted mandibular third molar.

Research design and methodology

Research method Quantitative

Type of study Experimental, double blinded, randomized comparaive study,

Study population Patient visiting department of oral and maxillofacial surgery in TUTH

Study site and its justification Large number of patients visit oral surgery department in TUTH.Most of them visit for surgical removal of impacted mandibular third molar and surgical extraction is commonly performed here.So oral and maxillofacial surgery OPD of TUTH will be ideal site for study as adequate sample size will be available without economic burden to the patient and investigator.

Sampling method Sampling method :Simple random sampling Randomisation will be done by random draw computer method Allocation concealment will be maintained using a sealed opaque envelope.

Sample size

Sample size will be calculated as; Sample size=2SD2(Z

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years
* No systemic illness and not taking any regular medications
* No signs of local inflammation
* Mesioangular and vertically impacted lower third molar
* Not under antibiotics for at least 3 days before surgery

Exclusion Criteria:

* With known systemic illness
* Those taking regular medications
* Presenting with pain and swelling at the time of surgery
* Impactions other than mesioangular and vertical impactions of lower third molar
* Under antibiotics within 3 days of surgical procedure
* Those having habit of cigarette smoking and females taking oral contraceptives

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
operative time taken for the surgical removal of impacted lower third molar | immediately after surgery
  The operative time taken will be recorded from the point of incision to the point of last suturing in terms of minutes.
postoperative pain Post operative pain which will be measured based on the questionnaires on defined post operative days | 1st postoperative day
  The postoperative pain will be measured by the visual analogue pain scale grading from 0 to 10 where score of 0 means no pain and 10 means maximum pain that can be felt by patient.
postoperative pain Post operative pain which will be measured based on the questionnaires on defined post operative days | 3rd postoperative day
  The postoperative pain will be measured by the visual analogue pain scale grading from 0 to 10 where score of 0 means no pain and 10 means maximum pain that can be felt by patient.
postoperative pain Post operative pain which will be measured based on the questionnaires on defined post operative days | 7th postoperative day
  The postoperative pain will be measured by the visual analogue pain scale grading from 0 to 10 where score of 0 means no pain and 10 means maximum pain that can be felt by patient.

SECONDARY OUTCOMES:
postoperative swelling | 1st postoperative day
  Measurement of edema will be done by using three facial lines ie. the tragus distance (point A) to the corner of the mouth (point C) , the tragus distance (point A) to pogonion (point D) and the angular distance (point E) to the lateral angle of the eye (point B). The distance between the three lines is measured in length and the average value is measured. Swelling will be measured as the difference between pre and post operative distance between these points in terms of millimeters.
postoperative swelling | 3rd postoperative day
  Measurement of edema will be done by using three facial lines ie. the tragus distance (point A) to the corner of the mouth (point C) , the tragus distance (point A) to pogonion (point D) and the angular distance (point E) to the lateral angle of the eye (point B). The distance between the three lines is measured in length and the average value is measured. Swelling will be measured as the difference between pre and post operative distance between these points in terms of millimeters.
postoperative swelling | 7th postoperative day
  Measurement of edema will be done by using three facial lines ie. the tragus distance (point A) to the corner of the mouth (point C) , the tragus distance (point A) to pogonion (point D) and the angular distance (point E) to the lateral angle of the eye (point B). The distance between the three lines is measured in length and the average value is measured. Swelling will be measured as the difference between pre and post operative distance between these points in terms of millimeters.
post operative trismus | 1st postoperative day
  Trismus will be measured as the difference in the distance between the incisal edge of the maxillary central incisor to the lower incisor in midline before and after surgery by using vernier caliper in terms of millimeters.
post operative trismus | 3rd postoperative day
  Trismus will be measured as the difference in the distance between the incisal edge of the maxillary central incisor to the lower incisor in midline before and after surgery by using vernier caliper in terms of millimeters.
post operative trismus | 7th postoperative day
  Trismus will be measured as the difference in the distance between the incisal edge of the maxillary central incisor to the lower incisor in midline before and after surgery by using vernier caliper in terms of millimeters.
dry socket | 3rd postoperative day
  The occurrence of dry socket will be observed by looking at whether there is an open alveolar bone area and the patient complaining of postoperative pain.
dry socket | 7th postoperative day
  The occurrence of dry socket will be observed by looking at whether there is an open alveolar bone area and the patient complaining of postoperative pain